CLINICAL TRIAL: NCT02627885
Title: Internet-based Cognitive Behavioral Therapy to Increase Function and Quality of Life for Patients With Parkinsons Disease
Brief Title: Internet-CBT for Parkinsons Disease
Acronym: Patrik
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Viktor Kaldo, Associate Professor (Docent), Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/1938-31/4
Record Dates: First submitted 2015-12-09; First posted 2015-12-11 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Parkinson Disease
Keywords: internet treatment; cognitive behavioral therapy; level of functioning; quality of life
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ICBT (Active Comparator): Internet-based CBT for Parkinsons Disease with therapist contact added to standard medical treatment
  Interventions: Behavioral: Internet-based CBT
- SMT (Other): Standard Medical Treatment for Parkinsons Disease only
  Interventions: Other: SMT

INTERVENTIONS:
Behavioral: Internet-based CBT — Through the use of CBT material at an Internet-platform, we aim for behavioral changes in the subjects to improve everyday level of functioning and quality of life.
  Arms: ICBT
Other: SMT — Standard Medical Treatment includes pharmacological management and other typical medical interventions for the patient group but no behavioural interventions
  Arms: SMT

SUMMARY:
The aim of the study is to investigate if an Internet-based psychological treatment based on principles from Cognitive Behavioral Therapy can increase function and quality of life for patients with Parkinson disease.

DETAILED DESCRIPTION:
The Internet-based Cognitive Behavioral Therapy (ICBT) will be given as an adjunct to the Standard Medical Treatment. ICBT will be compared to Standard Medical Treatment alone (SMT).

A secondary aim is make a preliminary evaluation of the ICBT-program with less and less active therapist support. It is hypothesized that both active treatments will be superior to SMT in improving quality of life and functioning and that ICBT with full therapist support will be superior to ICBT with lower level of therapist support.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Parkinson disease
* WSAS score of over 17
* Access to a internet connected device and a mobile phone capable of receiving SMS

Exclusion Criteria:

* Substance or alcohol abuse
* Psychotic Disorder or Bipolar disorder
* Other psychiatric disorder that requires immediate attention or hinders the offered ICBT treatment
* Practical obstacles such as difficulties using the technology required to participate in the study, not having the time to actively wok with the treatment, or having symptoms from Parkinson to severe to be able to actively participate in the study
* High suicide risk, defined as:
* 5 or 6 points on the question about Suicidal thoughts on the Montgomery-Asberg Depression Scale (MADRS)
* A standardized clinical interview on suicidal thoughts if the score on the above question is 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2015-12; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change (from baseline) in WSAS | Baseline, nine weekly measure while in treatment, then the primary endpoint is after 10 weeks of treatment (Post), and there will also be up to two follow-up (FU) measures within 3 years from treatment completion
  The Work and Social Adjustment Scale. Self-administered, measures impairment in functioning

SECONDARY OUTCOMES:
Change (from baseline) in IPAQ | Baseline, 5 weeks (Mid) 10 weeks (Post) and up to 2 (FU) measures
  International Physical Activity Questionnaire. Self-administered, measures physical activity
Change (from baseline) in SVAQ | Baseline, 5 weeks (Mid) 10 weeks (Post) and up to 2 (FU) measures
  Swedish Valued Activity Questionnaire. Self-administered, measures valued activities
Change (from baseline) in WHODAS-2 | Baseline, 10 weeks (Post) and up to 2 (FU) measures
  World Health Organization Disability Assessment Schedule 2 (12-item). Self-administered, measures disability
Change (from baseline) in PDQ-8 | Baseline, 10 weeks (Post) and up to 2 (FU) measures
  Parkinson's Disease Questionnaire-8. Self-administered, measures functioning and well-being patients with Parkinsons disease
Change (from baseline) in BBQ | Baseline, 10 weeks (Post) and up to 2 (FU) measures
  Brunnsviken Brief Quality of life scale. Self-administered, measures quality of life
Change (from baseline) in HADS | Baseline, 10 weeks (Post) and up to 2 (FU) measures
  The Hospital Anxiety and Depression Scale. Self-administered, measures anxiety and depression.
Change (from baseline) in ISI | Baseline, 10 weeks (Post) and up to 2 (FU) measures
  Insomnia Severity Index. Self-administered, measures insomnia and sleeping problems
Change (from baseline) in SSES6 | Baseline, 10 weeks (Post) and up to 2 (FU) measures
  Stanford Self-Efficacy for Managing Chronic Disease. Self-administered, measures self efficacy in relation to a chronic disease

OTHER OUTCOMES:
Adverse Events (self-rated) | 5 weeks (Mid) and 10 weeks (Post)
Adverse Events (therapist-rated) | 5 weeks (Mid) and 10 weeks (Post)
  Therapist use data from treatment to rate occurrences of Adverse events
Adverse Events (interviewer-rated) | 10 weeks (Post)
  Blind assessor asks about Adverse Events during whole treatment
Client Satisfaction | 10 weeks (Post)
  Client Satisfaction Questionnaire-8
Clinical Global Impression - Severity scale | 10 weeks (Post)
Clinical Global Impression - Improvement scale | 10 weeks (Post)
Use of other treatments | 10 weeks (Post)
  Use of other treatments during treatment period, self-rated

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Kaldo, Ph. D, Principal Investigator — Karolinska Institutet
Locations (1):
- Internetpsykiatrienehten (Internet Psychiatry Unit), Psykiatri Sydväst, SLSO Stockholm, Sweden, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kraepelien M, Schibbye R, Mansson K, Sundstrom C, Riggare S, Andersson G, Lindefors N, Svenningsson P, Kaldo V. Individually Tailored Internet-Based Cognitive-Behavioral Therapy for Daily Functioning in Patients with Parkinson's Disease: A Randomized Controlled Trial. J Parkinsons Dis. 2020;10(2):653-664. doi: 10.3233/JPD-191894. PMID 32176657